CLINICAL TRIAL: NCT06583252
Title: Effect of Multimodal Monitoring Cluster Management on Patients with Severe Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240707
Record Dates: First submitted 2024-09-01; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-06

CONDITIONS: Multimodal Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: multimodal monitoring cluster management — All patients will be monitored for baseline TCD at admission and at least once a day during treatment to assess changes in cerebral blood flow dynamics. Brain Oxygen Monitoring, Equipment & Frequency: Continuous monitoring of partial pressure of oxygen (PbtO2) in brain tissue using near-infrared spectroscopy (NIRS). qEEG monitoring，Frequency and timing of monitoring. Baseline monitoring: All patients will undergo a baseline qEEG test at the time of admission. Continuous monitoring: In the ICU, for critically ill patients, qEEG will be performed continuously to monitor changes in EEG activity in real time. Monitoring brain activity: qEEG is able to detect subtle changes in brain waves that can be used to assess brain functional status, such as EEG quiescence, abnormal electrical discharges (e.g., epileptiform activity), etc. Abnormal parameters: focus on abnormal rhythms (e.g., high-amplitude slow-wave activity), acute asymmetric activity, and epileptiform discharge.

SUMMARY:
Traumatic brain injury (TBI) is a serious global health problem, with about 27 million new cases each year. Severe head trauma can lead to intracranial hypertension and a range of complications such as cerebral edema and hypoxia of brain tissue. Intracranial pressure monitoring is key to modern TBI treatment, but this approach does not fully reflect all relevant pathophysiological changes. Multimodal monitoring allows for a more comprehensive assessment of the severity of TBI and guidance for individualized treatment to improve patient outcomes by integrating different monitoring methods. Although more research is needed to confirm its efficacy, multimodal monitoring has been recognized as an important clinical decision support tool in neuroscience intensive care. Future studies may further optimize this approach to monitoring and provide a more effective treatment strategy for patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

1.Age >18 years, 2.Diagnosis of an acute brain injury (ABI) due to TBI, 3.GCS with Eyes response = 1 (no eyes opening) and Motor score ≤5 (not following commands) at the admission to intensive care unit (ICU) or neuro-worsen-ing within the first 48 hours with no eye opening and the Motor score decreased to ≤5.

-

Exclusion Criteria:

1. Have had a major stroke before.
2. Pregnant or likely to become pregnant. 3 In the opinion of the treatment team, the decrease in GCS (Glasgow Coma Scale) score is solely due to intoxication, sedation, or extracranial injury.

4 Participants are unlikely to comply with all study procedures, including follow-up, in the opinion of the investigator.

5. Have an underlying medical condition with a life expectancy of less than 6 months.

6. There are pre-existing contraindications to MRI examination. 7 suffer devastating TBI, either progressing to brain death at the time of recruitment, or the treating medical team does not commit to continuous, comprehensive aggressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Score-Extended at 6 months | 6 months
  Glasgow Outcome Score-Extended at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No